CLINICAL TRIAL: NCT01021228
Title: Preconditioning is Indeed Protective
Brief Title: Preconditioning Volatile Anesthesia in Liver Surgery
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Slankamenac Ksenija, med. pract, Department of Visceral and Transplantation Surgery
Other Study IDs: StV 18-2008
Record Dates: First submitted 2009-11-25; First posted 2009-11-26 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2009-11

CONDITIONS: Anesthesia
Keywords: Liver resection; Continuous volatile anesthesia; Continuous intravenous anesthesia; Preconditioning volatile anesthesia; Comparing three groups of anesthesia during the liver surgery according to their benefit on liver and outcome.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- group1: continuous volatile anesthesia (sevoflurane) during the liver resection
- group2: continuous intravenous anesthesia (propofol) during the liver resection
- group3: preconditioning volatile anesthesia (sevoflurane) 30 minutes before ischemia (inflow occlusion)

SUMMARY:
The purpose of this study is to compare the impact and outcome of continuous volatile anesthesia to continuous intravenous anesthesia and to preconditioning volatile anesthesia in liver surgery.

DETAILED DESCRIPTION:
Comparing the impact and outcome of continuous volatile anesthesia to continuous intravenous anesthesia and to preconditioning volatile anesthesia in liver surgery.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* benign and malign disease
* any type of liver surgery
* inflow occlusion during the liver surgery

Exclusion Criteria:

* < 18 years
* participation on other interventional and treatment randomized controlled trials,
* trauma of the liver
* liver cirrhosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients were included undergoing any type of liver resection with inflow occlusion for benign as well as malign diseases between January first, 2005 and December 31, 2007 in a single tertiary care center
Sampling Method: Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2008-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
peak ALT and AST levels representing the ischemia-reperfusion injury | post-operative

SECONDARY OUTCOMES:
length of hospital stay, length of ICU stay, blood loss and morbidity (post-operative complications) | post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Ksenija Slankamenac, med. pract, Principal Investigator — Departement of Visceral and Transplantation
Locations (1):
- Universtiy Hospital of Zurich, Department of Visceral and Transplantation Surgery, Zurich, Canton of Zurich, Switzerland